CLINICAL TRIAL: NCT01712698
Title: Diffusion Tensor MRI to Assess Subacute Functional Outcomes in Patients With Acute Cervical Spinal Cord Injuries
Brief Title: Diffusion Tensor Imaging to Assess the Functional Outcomes of Adults With Cervical Spinal Cord Injuries
Status: Withdrawn | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: DTI; Washington University (Other: Washington University, St. Louis)
Record Dates: First submitted 2012-10-17; First posted 2012-10-23 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Cervical Spinal Cord Injury
Keywords: trauma; spinal cord injury; cervical spine
MeSH Terms: conditions — Wounds and Injuries; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cervical spinal cord injury: Those patients with an acute cervical spinal cord injury evaluated with DTI MRI

SUMMARY:
Acute changes in axial diffusivity will correlate with the severity of injury in patients that suffer an acute spinal cord injury.

DETAILED DESCRIPTION:
Diffusion tensor imaging (DTI) parameters will correlate with severity of spinal cord injury in SCI patients as seen in rodent models. We will test whether the quantitative decrease in axial (λ║) diffusivity (a biomarker of axonal injury), will predict long-term functional outcomes for patients with a SCI.

Specific Aim: To examine patients after an acute SCI using DTI and to correlate the extent of acute decrease in λ║ with the presenting ASIA motor score and long-term functional outcome of the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Cervical spinal cord injury
* physically and mentally willing to comply with imaging
* lives in immediate area with no plans to relocate

Exclusion Criteria:

* Associated moderate to severe head injury
* Active malignancy
* Previous spinal cord injury
* pregnancy
* inability to tolerate MRI scanning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a traumatic cervical spinal cord injury
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in AISA score | 24 months
  Patients will be followed for the duration of their hospital stay with clinical follow-up out to 2 years. ASIA scores will be correlated with admission DTI findings(Axial Diffusivity).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, School of Medicine, St Louis, Missouri, United States